CLINICAL TRIAL: NCT06182709
Title: Group Exposure Treatment: Feasibility of an Online Modeled Exposure in Spider Fearful Individuals
Brief Title: Feasibility of an Online Modeled Exposure in Spider Fearful Individuals
Acronym: OMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMEX_SPIDER
Record Dates: First submitted 2023-12-08; First posted 2023-12-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Spider Fear; Arachnophobia
MeSH Terms: conditions — Arachnophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- online modeled exposure + mental retrieval cue group exposure (Experimental): online modeled exposure training followed by group exposure training, including mental retrieval cue with five standardized exposure steps
  Interventions: Behavioral: online psychoeducation video + modeled exposure; Behavioral: group exposure; Behavioral: mental retrieval cue
- live modeled exposure + mental retrieval cue group exposure (Active Comparator): live modeled exposure training followed by group exposure training, including mental retrieval cue with five standardized exposure steps
  Interventions: Behavioral: live psychoeducation video + modeled exposure; Behavioral: group exposure; Behavioral: mental retrieval cue
- online modeled exposure + standardized group exposure (Active Comparator): online modeled exposure training followed by group exposure training with five standardized exposure steps
  Interventions: Behavioral: online psychoeducation video + modeled exposure; Behavioral: group exposure
- live modeled exposure + standardized group exposure (Active Comparator): live modeled exposure training followed by group exposure training with five standardized exposure steps
  Interventions: Behavioral: live psychoeducation video + modeled exposure; Behavioral: group exposure

INTERVENTIONS:
Behavioral: online psychoeducation video + modeled exposure — Participants will watch a short psychoeducation video online. This will be followed by a modeled exposure online. In this modeled exposure participants watch a film of an exposure treatment (about 45min) conducted with one participant and the therapist. The exposure training consists of five exposure steps (step 1: describing the spider, step 2: catching the spider with a glass, step 3: describing the spider, step 4: touching the spider with the dominant index finger, step 5: letting the spider walk on the participant hands; the following steps have to be repeated up to four times: 2,4,5).
  Arms: online modeled exposure + mental retrieval cue group exposure; online modeled exposure + standardized group exposure
Behavioral: live psychoeducation video + modeled exposure — Participants will watch a short psychoeducation video. This will be followed by a live modeled exposure. In this modeled exposure participants watch an exposure treatment (about 45min) conducted live with one participant and the therapist. The exposure training consists of five exposure steps (step 1: describing the spider, step 2: catching the spider with a glass, step 3: describing the spider, step 4: touching the spider with the dominant index finger, step 5: letting the spider walk on the participant hands; the following steps have to be repeated up to four times: 2,4,5).
  Arms: live modeled exposure + mental retrieval cue group exposure; live modeled exposure + standardized group exposure
Behavioral: group exposure — Exposure training in the group is conducted live (1 spider per participant, one therapist and co-trainers). In this group exposure participants complete exposure training (about 45 min) with five exposure steps (step 1: describing the spider, step 2: catching the spider with a glass, step 3: describing the spider, step 4: touching the spider with the dominant index finger, step 5: letting the spider walk on the participant hands; the following steps have to be repeated up to three times: 2,4,5).
Behavioral: mental retrieval cue — Before the group exposure, participants are asked to remember the modeled exposure they had observed the day before. Therefore, the participants are asked to recall the location where they have been during the modeled exposure and the reaction of the patient during the exposure (e.g., fear decline).
  Arms: live modeled exposure + mental retrieval cue group exposure; online modeled exposure + mental retrieval cue group exposure

SUMMARY:
The effectiveness of an optimized group exposure treatment is investigated in spider-fearful individuals. Participants will undergo an optimized standardized exposure treatment. After receiving information about the treatment and the phobic stimulus (spider) through a psychoeducation video, participants will observe an exposure treatment of another fearful person, either live or by watching a movie of an exposure treatment online. Subsequently, participants will undergo a live in vivo exposure treatment conducted in a group setting. The effectiveness of the treatment is measured by symptom improvement according to online behavioral avoidance tests and subjective ratings immediately after training and one week later.

DETAILED DESCRIPTION:
The treatment of various anxiety disorders often involves exposure therapy. However, a considerable number of patients do not benefit or experience a resurgence of anxiety following successful treatment. Vicarious safety learning (i.e., modeled exposure) presents a promising avenue to improve therapeutic outcome. Previous evidence indicates that vicarious safety learning can diminish previously acquired fear associations, thereby reducing behavioral avoidance. While single-session interventions have implemented modeled exposure, specific mechanisms of observational learning have not been extensively investigated. Due to high dropout rates in specific phobias, modeled exposure could be utilized as an additional treatment method, potentially yielding better outcomes trough additional learning experience.

This study aims to investigate the applicability of observational learning and its sustainability through mental retrieval cues. Specifically, the study is going to assess the feasibility of modeled exposure conveyed either live or online via video, offering a practical approach within a stepped-care framework. The modeled exposure treatment will be followed by a group exposure treatment to assess the influence of modeled exposure in spider-fearful individuals.

Physically healthy spider-fearful individuals will be either treated with an online or live modeled standardized exposure followed by a group exposure treatment. Half of the participants will receive a mental retrieval cue before the group exposure treatment one day after the modeled exposure treatment. The research aims to determine if long-term reduction of spider fear is achievable through online modeled exposure via video compared to in-person modeled exposure.

ELIGIBILITY:
Inclusion Criteria:

- Elevated score on Spider Phobia Questionnaire (SPQ) >= 17

Exclusion Criteria:

* Severe allergies to bees/spiders/insects
* Current psychiatric/psychotherapeutic treatment
* Past psychotherapeutic/psychiatric treatment due to anxiety problems
* Current or past psychotic symptoms
* Current suicidal intent
* Experience with exposure-based treatment
* Current psychopharmacological medication
* Severe respiratory, neurological or cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Spider Phobia Questionnaire (SPQ) | Change from baseline to immediately post treatment 1 (after modeled exposure), immediately post treatment 2 (group exposure) and follow-up (7 days after group exposure - post treatment 2)
  31-Item true/false questionnaire assessing symptoms of arachnophobia. Scores range from 0 to 31, with greater scores representing greater subjective fear of spiders, where lower scores reflect low subjective fear of spiders
Change in avoidance behavior (online virtual Behavioral Approach Task, vBATon) | Change from baseline to immediately post treatment 1 (after modeled exposure), immediately post treatment 2 (group exposure) and follow-up (7 days after group exposure - post treatment 2)
  Scores range from 0 ("participant refuses entering the room with the spider") to 12 ("participant holds the spider for at least 20 seconds")
Change in spider fear: Spider Anxiety Questionnaire (FSQ/SAF) | Change from baseline to immediately post treatment 1 (after modeled exposure), immediately post treatment 2 (group exposure) and follow-up (7 days after group exposure - post treatment 2)
  14-item questionnaire on a 7-point Likert-Scale (0 = "I don´t agree at all"; 6 = "I completely agree") to assess symptoms of arachnophobia. Total score can range from 0 to 98 Greater scores representing worse symptom severity of arachnophobia

SECONDARY OUTCOMES:
Change in spider phobia belief questionnaire (SBQ) | Change from baseline to immediately post treatment 1 (after modeled exposure), immediately post treatment 2 (group exposure) and follow-up (7 days after group exposure -- post treatment 2)
  Assessment of spider phobia dysfunctional beliefs; 48 items on a scale from 0% ("no approval") to 100% ("full approval"); higher scores indicate more dysfunctional beliefs about the danger of spiders and own coping abilities regarding spiders
Change in Spider Anxiety Screening (SAS) | Change from baseline to immediately post treatment 1 (after modeled exposure), immediately post treatment 2 (group exposure) and follow-up (7 days after group exposure- post treatment 2)
  Assessment of the four criteria for specific phobia (DSM-IV) with 4 items on a scale from 0 ("does not apply at all") to 6 ("fully applies"), Total score range: 0 to 24, higher scores indicating worse severity of symptoms of arachnophobia
Global success rating (GSR) | Change from immediately post treatment 1 (after modeled exposure) to immediately post-treatment 2 (after group exposure) and follow-up (7 days after group exposure- post treatment 2)
  Self-report measure of subjective state changes on a 7-likert scale from 1 ("much worse") to 7 ("much better")

OTHER OUTCOMES:
Anxiety Sensitivity (ASI-3) | baseline
  Self-report measure of anxiety-related body symptoms (i.e. anxiety sensitivity) with 18 items on a scale from 0 ("does not apply at all") to 4 ("fully applies"). Total score can range from 0 to 72; higher scores indicate worse anxiety sensitivity
Depression, Anxiety and Stress Scale (DASS) | baseline
  Self-report measure of main symptoms of depression, anxiety, and stress, 21 items on a 4-point severity/frequency scale from 0 ("didn´t apply to me at all") to 4 ("applied very much to me, or most of the time"). Total score can range from 0 to 84, higher scores indicate higher symptom severity
Group Entitativity Measure-Group Therapy (GEM-GP) | immediately post-treatment 2 (after group exposure)
  Single item visual analogue scale to measure group cohesion, scale can range from 1 to 6, higher scores indicate higher group cohesion
Group Climate Questionnaire (GCQ-S) | immediately post-treatment 2 (after group exposure)
  Self-report measure assessing perception of group atmosphere on 12 items rated on a 7-point Likert-scale (0 = "not at all" to 6 = "very much/extremely")
Muenster Epistemic Trustworthiness Inventory (METI) | Change from immediately post treatment 1 (after modeled exposure) to immediately post-treatment 2 (after group exposure)
  Self-report measure of epistemic trustworthiness, consisting of 14 antonyms on a 7-point scale, higher scales indicate higher epistemic trust
Intolerance of uncertainty (IUS-12) | baseline
  Self-report measure to assess uncertainty intolerance with 12 items on a 5-point Likert-scale from 1 ("not at all characteristics of me") to 5 ("very characteristic of me"), higher scores indicate greater uncertainty intolerance
Positive mental health Scale (PMH) | baseline
  Self-report measure assessing emotional and psychological aspects of wellbeing with 9 items rated on a scale from 0 ("do not agree") to 3 ("agree"), score can range from 0 to 27, higher scores indicate greater wellbeing
Interpersonal Reactivity Index (IRI) | baseline
  Self-report measure to assess empathy with 16 Items on a scale from 0 ("never") to 4 ("always"), score can range from 0 to 66, higher scores indicate greater empathy
State-Trait Anxiety Inventory - Trait (STAI-T) | baseline
  Self-report measure of general anxiety with 20 Items (range from 1 = "almost never" to 4 = "nearly always"), Score range from 20 (no anxiety) to 80 (high anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane A. Melzig, PhD, Principal Investigator — Philipps University Marburg; Jana Gessner, M.Sc., Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craske MG, Treanor M, Conway CC, Zbozinek T, Vervliet B. Maximizing exposure therapy: an inhibitory learning approach. Behav Res Ther. 2014 Jul;58:10-23. doi: 10.1016/j.brat.2014.04.006. Epub 2014 May 9. PMID 24864005
- [Background] Golkar A, Selbing I, Flygare O, Ohman A, Olsson A. Other people as means to a safe end: vicarious extinction blocks the return of learned fear. Psychol Sci. 2013 Nov 1;24(11):2182-90. doi: 10.1177/0956797613489890. Epub 2013 Sep 10. PMID 24022651
- [Background] Ost LG, Ferebee I, Furmark T. One-session group therapy of spider phobia: direct versus indirect treatments. Behav Res Ther. 1997 Aug;35(8):721-32. doi: 10.1016/s0005-7967(97)00028-4. PMID 9256515
- [Background] Mystkowski JL, Craske MG, Echiverri AM, Labus JS. Mental reinstatement of context and return of fear in spider-fearful participants. Behav Ther. 2006 Mar;37(1):49-60. doi: 10.1016/j.beth.2005.04.001. Epub 2006 Feb 24. PMID 16942960
- [Background] Olsson A, Phelps EA. Social learning of fear. Nat Neurosci. 2007 Sep;10(9):1095-102. doi: 10.1038/nn1968. PMID 17726475
- [Background] Wannemueller A, Appelbaum D, Kuppers M, Matten A, Teismann T, Adolph D, Margraf J. Large Group Exposure Treatment: a Feasibility Study in Highly Spider Fearful Individuals. Front Psychol. 2016 Aug 9;7:1183. doi: 10.3389/fpsyg.2016.01183. eCollection 2016. PMID 27555830